CLINICAL TRIAL: NCT04850612
Title: Defining Core Outcomes and Data Elements (CODE) in Chronic Subdural
Brief Title: Defining Core Outcomes and Data Elements (CODE) in Chronic Subdural Haematoma
Acronym: CODE-CSDH
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Erasmus Medical Center (Other); Université de Sherbrooke (Other); Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Ellie Edlmann, Clinical Lecturer in Neurosurgery, University Hospital Plymouth NHS Trust
Other Study IDs: CA_2020-21-303
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Chronic Subdural Hematoma
Keywords: head injury; core outcome set; elderly
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Craniocerebral Trauma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthcare professionals and researchers (HCPR): All researchers and healthcare professionals involved in the management of patients with CSDH
  Interventions: Other: Survey
- Patients and carers: Patients who have previously had a diagnosis of CSDH, and their carers
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Delphi Survey on core outcomes, CSDH definition and data elements

SUMMARY:
This study is aimed at improving reporting in Chronic Subdural Haematoma (CSDH) research studies, through development of a standardised Core Outcome Set (COS), a unified CSDH Definition and set of Data Elements (DE) for reporting.

The study design includes a Delphi survey process from two main stakeholder groups: Health-Care Professionals or Researchers (HCPR) and Patients or carers. HCPR, patients and carers will all be invited to complete the survey on the COS, only the HCPR survey will include questions on definition and DE. Results of the Delphi Survey will be discussed at a final consensus meeting before results are confirmed and published.

DETAILED DESCRIPTION:
Chronic subdural haematoma (CSDH) is a collection of blood and fluid surrounded by membranes that accumulates on the brain surface over weeks to months. It predominately affects older people and often has a delayed association with a preceding head trauma.

There has been significant growth in the number of CSDH publications in recent years mirroring progress in potential management options but there is wide variation in how and when patient outcome is measured amongst studies. Much could be gained by agreeing a minimum set of standardized outcomes that should be measured and reported in all CSDH studies, known as a Core Outcome Set (COS).

The overall study design includes a Delphi survey process.This is a process whereby all outcomes and data elements from the CSDH literature and expert opinion are presented to a large group of patients, carers and HCPR via a survey. Each survey participant has the opportunity to rank the elements and outcomes in levels of importance to them, and the survey is then repeated including presentation of the results from the first round, in order to attempt to gain agreement between participants on what is important. All elements are then reviewed at a final "consensus" meeting

ELIGIBILITY:
Inclusion Criteria:

All invited participants who provide consent to take part in 2 rounds of survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare Professionals, Researchers, patients and carers.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
CSDH Core Outcome Set (COS) | 3 months
  Definition of a Core Outcome Set (COS) for reporting in all future CSDH studies through a Delphi survey process including all relevant stakeholders.

SECONDARY OUTCOMES:
CSDH Definition and Data Elements | 3 months
  Identify a unified CSDH definition and data elements (DE) for reporting in future CSDH studies, through a Delphi survey process including healthcare profession and research (HCPR) stakeholders.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Protocol submitted for open publication prior to commencing study. Final study report will be published at end of study including full anonymised survey responses.